CLINICAL TRIAL: NCT01246752
Title: Randomised Trial on Allogeneic Haematopoietic Stem Cell Transplantation in Patients Under the Age of 60 Years With Acute Myeloid Leukemia of Intermediate Risk in First Complete Remission and a Matched Sibling or Unrelated Donor (ETAL-1)
Brief Title: Haematopoietic Stem Cell Transplantation (HSCT) in Comparison to Conventional Consolidation Therapy for Patients With Acute Myeloid Leukemia (AML) (Intermediate Risk) </= 60y. After First CR
Acronym: AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: decreased recrucial rate as the likelihood of achieving the envisioned patient number in a realistic time-frame was very low.
Sponsor: University Hospital Carl Gustav Carus (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-ETAL-1-045
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML, Leukemia; Acute Myeloid Leukemia; HSCT; Stem Cell Transplantation; Tx; Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Consolidation Chemotherapy; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Stem Cell Transplantation (Experimental): Patients receive an allogenic stem cell transplantation from an HLA-matched unrelated or related donor
  Interventions: Biological: Human Stem Cell Transplantation
- Consolidating Chemotherapy (Active Comparator): Patients receive a standard chemotherapy as consolidation therapy
  Interventions: Drug: Consolidation chemotherapy, i.e. High-dose Cytarabine (HiDAC)

INTERVENTIONS:
Biological: Human Stem Cell Transplantation — Human allogenic stem cells
  Arms: Human Stem Cell Transplantation
Drug: Consolidation chemotherapy, i.e. High-dose Cytarabine (HiDAC) — Consolidation chemotherapy, recommended regimen: HiDAC = 3 x 2g/sqm BID on days 1,3,5
  Arms: Consolidating Chemotherapy

SUMMARY:
Hematopoietic stem cell transplantation in patients with newly diagnosed AML ≤60 years of age in intermediate risk, after first complete response in comparison to standard consolidation chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* AML in first remission
* cytological standard risk, i.e. karyotype not listed under exclusion criteria
* Identification of HLA-identical sibling or HLA-compatible related or unrelated donor (9/10 HLA-alleles matched, high resolution typing for HLA-A, B, Cw, DRB1 and DQB1)
* age: 18 - 60 years
* medically fit for allogeneic stem cell transplantation
* CR / CRi after induction therapy

Exclusion Criteria:

* core-binding factor leukemia (t(8;21), inv16)
* acute promyelocytic leukemia (t(15;17)
* complex aberrant karyotype
* karyotypes: -7; -5; del5q; t(3;3); t(6;11), t(6;9), 11q aberrations, trisomy 8 ± one single additional aberration
* pregnancy / nursing
* non-compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2011-02-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Percent of Patients alive after 4 years (Overall Survival) | 4 years
  The status of each patient alive/not alive is surveyed every 3 months in year 1+2 and every 6 months in year 3+4 after randomisation.

SECONDARY OUTCOMES:
Disease-free survival | 4 years
Cumulative incidence of relapse | 4 years
Cumulative incidence of non-relapse mortality | 4 years
Quality of life assessed by questionnaires | 4 years
  Scores assessed by validated questionnaires (8 subscales: physical function, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bornhaeuser, Prof. (MD), Principal Investigator — Universitätsklinikum Dresden, Medizinische Klinik und Poliklinik I, Germany
Locations (19):
- Germany (19):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - University Hospital Carl Gustav Carus, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen - Westdeutsches Tumorzentrum, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Klinikum der Johann-Wolfgang-Goethe Universität, Frankfurt am Main
  - Universitätsklinikum Halle, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Universitaetsklinikum Leipzig - AöR, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Klinikum der LMU Universität - Campus Großhadern, München
  - Universitätsklinikum Münster, Münster
  - Städtisches Klinikum Nord, Nuremberg
  - Ernst-von-Bergmann-Klinikum Potsdam, Potsdam
  - Robert-Bosch-Krankenhaus, Stuttgart

REFERENCES:
- [Derived] Bornhauser M, Schliemann C, Schetelig J, Rollig C, Kramer M, Glass B, Platzbecker U, Burchert A, Hanel M, Muller LP, Klein S, Bug G, Beelen D, Rosler W, Schafer-Eckart K, Schmid C, Jost E, Lenz G, Tischer J, Spiekermann K, Pfirrmann M, Serve H, Stolzel F, Alakel N, Middeke JM, Thiede C, Ehninger G, Berdel WE, Stelljes M. Allogeneic Hematopoietic Cell Transplantation vs Standard Consolidation Chemotherapy in Patients With Intermediate-Risk Acute Myeloid Leukemia: A Randomized Clinical Trial. JAMA Oncol. 2023 Apr 1;9(4):519-526. doi: 10.1001/jamaoncol.2022.7605. PMID 36757706
- See also: Study Alliance Leukemia (coordinating study group) — http://www.sal-aml.org